CLINICAL TRIAL: NCT02757235
Title: The Swedish Study of Irrigation Fluid Temperature in the Evacuation of Chronic Subdural Hematoma - A Multicenter Randomised Controlled Trial
Brief Title: The Swedish Study of Irrigation Fluid Temperature in the Evacuation of Chronic Subdural Hematoma
Acronym: SIC!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Bartley, MD, neurosurgical resident, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIC01
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma; irrigation; recurrence; burr hole evacuation; temperature
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irrigation fluid of body temperature (Active Comparator): During burr hole evacuation of the chronic subdural hematoma the irrigation fluid used will be of body temperature (approximately 37 degrees Celsius)
  Interventions: Procedure: Irrigation fluid of body temperature
- Irrigation fluid of room temperature (Active Comparator): During burr hole evacuation of the chronic subdural hematoma the irrigation fluid used will be of room temperature (approximately 22 degrees Celsius)
  Interventions: Procedure: Irrigation fluid of room temperature

INTERVENTIONS:
Procedure: Irrigation fluid of body temperature — Irrigation fluid of body temperature will be used during burr hole evacuation of chronic subdural hematoma
  Arms: Irrigation fluid of body temperature
Procedure: Irrigation fluid of room temperature — Irrigation fluid of room temperature will be used during burr hole evacuation of chronic subdural hematoma.
  Arms: Irrigation fluid of room temperature

SUMMARY:
The study will be a multicenter randomised controlled trial of the use of irrigation fluid of body temperature versus irrigation fluid of room temperature during burr hole evacuation of chronic subdural hematoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic subdural hematoma requiring burr hole evacuation.
* Patients older than 18 years of age.

Exclusion Criteria:

* Chronic subdural hematoma requiring surgical treatment other than burr hole evacuation.
* Chronic subdural hematoma in a patient with an intracranial arachnoidal cyst.
* Chronic subdural hematoma in a patient with a Cerebro Spinal Fluid-shunt.
* Patients who have undergone intracranial surgery before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2016-03; Primary Completion 2020-10 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 6 months
  Recurrences requiring repeat surgery during a 6-month follow up period

SECONDARY OUTCOMES:
Mortality | 6 months
  The proportion deceased at a given time during the 6 month follow up.
Complications related to the surgery | 6 months
  Complications will be assessed using the Landriel Ibanez classification modelThis model grades complications in 4 grades (Grade 1: no invasive treatment required; Grade 2: invasive treatment required, but not intensive care; Grade 3: invasive treatment required and intensive care; Grade 4: death).
Health related quality of life | 6 months
  A standardised instrument, EuroQoL 5D-3L, will be used as a generic measure of health related quality of life. The questionnaire contains 5 questions in different domains.

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir Jakola, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Department of neurosurgery; Niklas Marklund, MD, Phd, Principal Investigator — Akademiska University Hospital, Department of neurosurgery; Jimmy Sundblom, MD, Phd, Principal Investigator — Akademiska University Hospital, Department of neurosurgery; Jiri Bartek, MD, Principal Investigator — Karolinska University Hospital, Department of neurosurgery; Andreas Bartley, MD, Principal Investigator — Sahlgrenska University Hospital, Department of neurosurgery; Magnus Tisell, MD, PhD, Study Director — Sahlgrenska Universtiy Hospital, Department of neurosurgery; Petter Förander, MD, PhD, Principal Investigator — Karolinska University Hospital, Department of neurosurgery
Locations (3):
- Sweden (3):
  - Sahlgrenska Universtity Hospital, Department of neurosurgery, Sweden, Gothenburg
  - Karolinska University Hospital, Department of neurosurgery, Sweden, Solna
  - Uppsala University Hospital, Department of neurosurgery, Sweden, Uppsala

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bartley A, Bartek J Jr, Jakola AS, Sundblom J, Falt M, Forander P, Marklund N, Tisell M. Effect of Irrigation Fluid Temperature on Recurrence in the Evacuation of Chronic Subdural Hematoma: A Randomized Clinical Trial. JAMA Neurol. 2023 Jan 1;80(1):58-63. doi: 10.1001/jamaneurol.2022.4133. PMID 36409480
- [Derived] Bartley A, Jakola AS, Bartek J Jr, Sundblom J, Forander P, Marklund N, Tisell M. The Swedish study of Irrigation-fluid temperature in the evacuation of Chronic subdural hematoma (SIC!): study protocol for a multicenter randomized controlled trial. Trials. 2017 Oct 11;18(1):471. doi: 10.1186/s13063-017-2194-y. PMID 29021000